CLINICAL TRIAL: NCT02718742
Title: Maintenance Nab-Paclitaxel After Cisplatin-Based Neoadjuvant Chemotherapy in Patients With High Risk Bladder Cancer
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation After Cisplatin-Based Chemotherapy and Surgery in Treating Patients With High-Risk Bladder Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1551; NCI-2016-00133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1551 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2016-02-10; First posted 2016-03-24 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Recurrent Bladder Urothelial Carcinoma; Stage IV Bladder Urothelial Carcinoma
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nab-paclitaxel) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; nab-paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; protein-bound paclitaxel
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well paclitaxel albumin-stabilized nanoparticle formulation maintenance therapy works after cisplatin-based chemotherapy and surgery in treating patients with high-risk bladder cancer. Maintenance therapy, such as paclitaxel albumin-stabilized nanoparticle formulation, can help keep cancer from coming back after it has disappeared following initial chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 6-month progression-free survival (PFS) rate in patients with high risk urothelial carcinoma treated with cisplatin-based neoadjuvant chemotherapy followed by curative intent cystectomy receiving maintenance therapy with paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel).

SECONDARY OBJECTIVES:

I. To evaluate overall survival (OS), time to progression and duration of response in patients treated with cisplatin-based neoadjuvant chemotherapy followed by curative intent cystectomy receiving maintenance therapy with nab-paclitaxel.

II. To evaluate the adverse events associated with use of single agent nab-paclitaxel (Abraxane®) in patients with high risk urothelial carcinoma receiving maintenance therapy III. To evaluate Health Related Quality of life (HRQoL) as assessed by the European Organization for Research and Treatment of Care (EORTC) QLQ-C30.

TERTIARY OBJECTIVES:

I. To determine the presence of circulating tumor cells (CTC) in high risk patients with urothelial carcinoma prior to initiation of maintenance therapy (baseline) and after nab-paclitaxel exposure (at cycles 2, 4).

OUTLINE:

Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of urothelial carcinoma and high risk residual disease after neoadjuvant chemotherapy (NAC) and cystectomy as defined by post-operative pathological pT4 or N1-3 disease, or progressive disease during NAC (NAC include methotrexate, vinblastin, doxorubicin and cisplatin [MVAC], dose dense MVAC, gemcitabine cisplatin, or gemcitabine carboplatin); minor histologic variants (< 50%) are acceptable if urothelial carcinoma is predominant variant
* Post-operative computed tomography (CT) scan of the chest, abdomen, and pelvis =< 30 days prior to registration demonstrating no evidence of residual or recurrent malignancy
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x upper limit of normal (ULN)
* Creatinine =< 1.5 mg/dL or creatinine clearance >= 40mL/mon (using Cockcroft-Gault formula)
* Females of child-bearing potential, defined as a sexually mature woman who (1) has not undergone hysterectomy or bilateral oophorectomy or (2) has not been naturally postmenopausal for at least 24 consecutive months must:

  * Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting intraperitoneal (IP) therapy (including dose interruptions), and while on study medication or for a longer period if required by local regulations following the last dose of IP
  * Negative serum pregnancy test done =< 7 days prior to registration and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy; this applies even if the subject practices true abstinence from heterosexual contact
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during those interruptions and for 6 months following IP discontinuation, even if he has undergone a successful vasectomy
* Patients must have =< grade 2 pre-existing peripheral neuropathy (per Common Terminology Criteria for Adverse Events [CTCAE] v4.0)
* Ability to complete questionnaire(s), in English, by themselves or with assistance
* Provide informed written consent
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Radiographic evidence measurable of residual or metastatic disease after surgery
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects to a developing fetus or nursing child:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration except for locally curable cancers that have been in apparently cured, such as basal or squamous cell skin cancer, prostate cancer without evidence of prostate-specific antigen (PSA) progression or carcinoma in situ such as the following: gastric, cervix, colon, melanoma or breast for example
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Pure small cell histologic variant or other pure non-urothelial carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of progression-free survivors assessed by Response Evaluation Criteria for Solid Tumors (RECIST) | 6 months
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated using the approach of Duffy and Santner. Additionally, if some patients are lost to follow-up not having been observed for at least 6 months, an estimate and confidence interval for the 6-month progression-free survival rate incorporating censoring will be computed using the method of Kaplan-Meier (1958).

SECONDARY OUTCOMES:
Duration of response assessed by RECIST | From the date at which the patient's earliest best objective status is first noted to be at least a partial response or better to the earliest date progression is documented
  The distribution of duration of response will be estimated using the method of Kaplan-Meier (1958).
Frequency and severity of observed adverse effects assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) | Up to 2 years
Overall survival (OS) | From the date of registration to the event of death due to any cause, up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier (1958).
Quality of life assessed using the EORTC QLQ-C30 | At baseline, before each chemotherapy cycle, at end of treatment and at 3 and 6 month observation visits
  28 of the 30 items are measured on a 1-4 scale (1=not at all; 4=very much) with the remaining two items (overall health and overall quality of life) scored on a 1-7 numeric analogue scale (1=very poor; 7=excellent). The recall period for the EORTC QLQ-C30 is one week.
Time to disease progression assessed by RECIST | From the date of registration to the earliest date of documentation of disease progression, up to 2 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier (1958).

CONTACTS AND LOCATIONS:
Overall Officials: Estrella Carballido, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States